CLINICAL TRIAL: NCT05605418
Title: Study of a Comprehensive Intelligent Hypertension managEment SyStem (CHESS) Evaluation in Primary Health Care Settings
Brief Title: Study of a Comprehensive Intelligent Hypertension managEment SyStem
Acronym: CHESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-GSP-GG-21
Record Dates: First submitted 2022-10-27; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Hypertension
Keywords: Hypertension; Digital intervention; Ambulatory blood pressure; Home blood pressure monitoring; Cluster randomized controlled trial
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHESS intervention (Experimental): Physicians and patients at the intervention group will receive training and support on the use of the multi-faceted CHESS system.
  Interventions: Behavioral: CHESS intervention
- Control (No Intervention): After site randomization, physicians at the control sites will manage their patients by usual care at hypertension clinics.

INTERVENTIONS:
Behavioral: CHESS intervention — The multi-faceted CHESS intervention includes: (1) home blood pressure monitoring (HBPM) for patients, and the data will be uploaded to central electronic health records (EHR) automatically; (2) a Smart Reminder and Alert System (SRAS) to send educational messages and reminders to support patients on HBPM, improve blood pressure medication adherence and lifestyle modification; (3) a decision support system (DSS) to provide physicians with antihypertensive medications prescriptions and referral recommendations; (4) regular quality assessment reports will be provided to health care providers automatically to improve the quality of hypertension management at PHC level.
  Arms: CHESS intervention

SUMMARY:
This cluster randomized controlled trial aims to evaluate the efficacy of a comprehensive intelligent hypertension management system (CHESS) in blood pressure lowering in primary health care (PHC) settings of China.

DETAILED DESCRIPTION:
The trial aims to investigate the efficacy of a comprehensive digital intervention for hypertension treatment in cluster clinics. 40 PHC centers will be selected from different areas in China, and eligible patients being screened consecutively in each site, then all PHC centers will be randomized into intervention group and control group. The physicians and patients from the 20 intervention sites will receive training and support on the use of the CHESS system, and the control group will continue to receive usual care. The multi-faceted CHESS intervention includes: (1) home blood pressure monitoring (HBPM) for patients, and the data will be uploaded to central electronic health records (EHR) automatically; (2) a Smart Reminder and Alert System (SRAS) to send educational messages and reminders to support patients on HBPM, improve blood pressure medication adherence and lifestyle modification; (3) a decision support system (DSS) to provide physicians with antihypertensive medications prescriptions and referral recommendations; (4) regular quality assessment reports will be provided to health care providers automatically to improve the quality of hypertension management at PHC level. All participants will be asked to attend the clinic at least once every 3 months, and be followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria for Sites:

1. An electronic data collection system is routinely used at the clinic for hypertension management in PHC sites, and the distance between sites must be >2km;
2. At least one drug of each of the five classes of recommended antihypertensive medications is available at the clinic:

   * A: Angiotensin-converting enzyme inhibitors (ACEI; e.g., captopril or enalapril);
   * A: Angiotensin receptor blockers (ARB; e.g., losartan or valsartan)
   * B: β-blockers (e.g., atenolol, metoprolol, or bisoprolol)
   * C: Calcium antagonists (e.g., nitrendipine, nifedipine, or amlodipine)
   * D: Diuretics (e.g., hydrochlorothiazide, indapamide, or indapamide SR tablets)
3. Has an outpatient clinic for hypertension treatment and staff are willing to take part in the study.

Inclusion Criteria for Participants:

1. Age ≥35 years and <80 years
2. Local resident of the community/township who attends the PHC clinic for hypertension management, and will not travel for more than 3 months during the study period;
3. Established diagnosis of essential hypertension, with uncontrolled BP before randomization (defined as office BP≥140/90mmHg, and 24-hour ambulatory BP≥130/80mmHg);
4. Own and be able to use a smartphone daily;
5. Be willing to participate in the study and sign the informed consent.

Exclusion Criteria for participants:

1. Physician-diagnosed or suspected secondary hypertension (e.g. hypertension caused by renal disease, renal artery stenosis, aortic stenosis, primary aldosteronism, pheochromocytoma/paraganglioma, Cushing's syndrome, thyroid dysfunction, intracranial disease, drug- induced, or rare monogenic genetic disease), or the presence of other structural heart diseases, such as aortic insufficiency, hypertrophic cardiomyopathy, or congenital heart disease;
2. Office or ambulatory SBP≥180 mmHg and/or DBP≥110 mmHg before randomization;
3. Physician-diagnosed atrial fibrillation;
4. Physician-diagnosed CKD, estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 (if serum creatinine is available), or currently on dialysis treatment;
5. Physician-diagnosed hepatic dysfunction, or ALT≥ 2*ULN;
6. Currently at the unstable or terminal stage of any disease (e.g. new- onset cardiovascular and cerebrovascular diseases occurred within 3 months, malignant tumors);
7. Intolerance to at least two classes of antihypertensive medications among A, B, C or D;
8. Currently taking 3 or more antihypertensive drugs;
9. The subject is pregnant or breastfeeding, or planning to become pregnant or breastfeeding during the study period;
10. Have communication or cognitive disorders;
11. Be unwilling to take antihypertensive drugs, or assumed poor adherence to treatment;
12. The subject is participating in other clinical trials at the moment.

Ages: 35 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in 24-hour ambulatory SBP from baseline to 12-month follow up; | Baseline; 12 months
  The investigators will measure the change in 24-h ambulatory SBP from baseline to 12 months.

SECONDARY OUTCOMES:
Mean changes in 24-hour ambulatory DBP from baseline to 12-month; | Baseline; 12 months
  The investigators will measure the change in 24-h ambulatory DBP from baseline to 12 months.
Mean changes in office SBP from baseline to 12-month; | Baseline; 12 months
  Patient's office SBP will be measured at hypertension clinics.
Mean changes in office DBP from baseline to 12-month; | Baseline; 12 months
  Patient's office DBP will be measured at hypertension clinics.
Proportion of patients with office BP under control at 12-month; | Baseline; 12 months
  Office BP under control is defined as blood pressure <130/80 mmHg at hypertension clinic.
Proportion of patients with 24-hour ambulatory BP under control (<130/80 mmHg) at 12-month; | Baseline; 12 months
  Ambulatory BP under control is defined as mean ambulatory BP <130/80 mmHg.
Mean changes in 24-hour ABPM heart rate from baseline to 12-month; | Baseline; 12 months
  The investigators will measure the change in 24-h ambulatory heart rate from baseline to 12 months.
Proportion of hypertension visits during which inappropriate antihypertensive treatment is prescribed; | Baseline; 12 months
  Inappropriate antihypertensive treatment is defined as a prescription incompliant with the pre-specified guideline-based recommendations. Antihypertensive treatment prescriptions will be measured and obtained through questionnaire and medical records information and be compared with decision support system recommendations automatically.
Change in patients' medication adherence of antihypertensive drugs; | Baseline; 12 months
  The investigators will measure patients medication adherence using information collected in questionnaire at baseline and 12 month follow up visits.

OTHER OUTCOMES:
Mean changes in ambulatory daytime SBP from baseline to 12-month; | Baseline; 12 months
  Ambulatory daytime SBP will be measured according to 24-hour ABPM.
Mean changes in ambulatory daytime DBP from baseline to 12-month; | Baseline; 12 months
  Ambulatory daytime DBP will be measured according to 24-hour ABPM.
Mean changes in ambulatory nighttime SBP from baseline to 12-month; | Baseline; 12 months
  Ambulatory nighttime SBP will be measured according to 24-hour ABPM.
Mean changes in ambulatory nighttime DBP from baseline to 12-month; | Baseline; 12 months
  Ambulatory nighttime DBP will be measured according to 24-hour ABPM.
Mean changes in BMI from baseline to 12-month; | Baseline; 12 months
  BMI will be measured by dividing weight in kilograms by height in metres squared.
Changes in physical activity level from baseline to 12-month; | Baseline; 12 months
  We will measure the change in self-reported physical activity scale through questionnaire from baseline to 12 months.
Changes in smoking proportions from baseline to 12-month; | Baseline; 12 months
  We will measure the change in self-reported smoking status through questionnaire from baseline to 12 months.
Proportions of patients with major cardiovascular events during follow-up period. | Baseline; 12 months
  Major cardiovascular events are defined as cardiovascular death, non-fatal myocardial infarction, non-fatal stroke, and hospitalization for heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, PhD, Principal Investigator — National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, National Center for Cardiovascular Diseases, Beijing, China

REFERENCES:
- [Derived] Zhang H, Huo X, Ren L, Lu J, Li J, Zheng X, Liu J, Ma W, Yuan J, Diao X, Wu C, Zhang X, Wang J, Zhao W, Hu S. Design and rationale of the Comprehensive intelligent Hypertension managEment SyStem (CHESS) evaluation study: A cluster randomized controlled trial for hypertension management in primary care. Am Heart J. 2024 Jul;273:90-101. doi: 10.1016/j.ahj.2024.03.018. Epub 2024 Apr 2. PMID 38575049